CLINICAL TRIAL: NCT01390896
Title: Special Drug Use Investigation for ARIXTRA (Fondaparinux) Abdominal General Surgery
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112797
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fondaparinux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed fondaparinux: Patients undergoing general surgery of the lower limb at high risk for venous thromboembolism
  Interventions: Drug: Fondaparinux Sodium

INTERVENTIONS:
Drug: Fondaparinux Sodium

SUMMARY:
The purpose of this study is to collect and assess information on safety and efficacy of fondaparinux in patients undergoing general surgery of the lower limb at high risk of developing venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general surgery of the lower limb at high risk for venous thromboembolism

Exclusion Criteria:

* Patients with a history of hypersensitivity to the ingredients of fondaparinux
* Patients with bleeding (bleeding in important organs, sucn as retroperitoneal bleed)
* Patients with acute bacterial endocarditis
* Patients with severe renal impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients undergoing general surgery of the lower limb at high risk for venous thromboembolism
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects undergoing general surgery of the lower limb treated with fondaparinux | 1 month
Presence of absence of venous thromboembolism after treatment of fondaparinux | 1 month
Occurrence of adverse events of bleeding | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline